CLINICAL TRIAL: NCT01350401
Title: Phase I/II Study to Assess the Safety and Activity of Enhanced TCR Transduced Autologous T Cells in Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP 01611
Record Dates: First submitted 2011-05-02; First posted 2011-05-09 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Melanoma
Keywords: Melanoma; Cell Therapy; T Cell Therapy; NY-ESO-1; Immuno-oncology; Metastatic; Previously treated; T Cell Receptor
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NY-ESO-1/LAGE-1 and HLA-A*02 Positive Subjects (Experimental)
  Interventions: Genetic: Autologous genetically modified T cells, NY-ESO-1ᶜ²⁵⁹T

INTERVENTIONS:
Genetic: Autologous genetically modified T cells, NY-ESO-1ᶜ²⁵⁹T — Cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T

SUMMARY:
The purpose of this early (phase I/II) clinical trial is to assess the effects (both good and bad) of genetically modified T cells after chemotherapy on your cancer and general health.

DETAILED DESCRIPTION:
Purpose of this study is to evaluate the safety and tolerability of autologous genetically modified T cells. Genetic material is transferred into the subject's previously harvested autologous T cells to redirect them to target melanoma cells rather than their usual target. Study subjects must have histologically or cytologically melanoma stage 3/4 and their tumor must express HLA Class 1 allele HLA-A*0201 for NY-ESO-1/LAGE. Subjects must also have measureable disease on study entry, as defined by at least one lesion that can be measured in at least one dimension >= 10mm with spiral CT scan.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically or cytologically confirmed melanoma stage III/IV, unresectable
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with spiral CT scan
* One prior cytotoxic therapy for the treatment of metastatic disease is allowed. Unlimited regimens using biological agents (vaccines), immunotherapy, or targeted agents is permitted. For example, BRAF inhibitors and ipilimumab are permitted. Patients must have fully recovered from the acute toxicities related to any prior therapy. Prior therapy must be completed ≥28 days before the first dose of cyclophosphamide.
* Age ≥18
* Life expectancy of greater than 3 months
* ECOG performance status ≤ 1

Patients must have normal organ and marrow function as defined below:

* Leukocytes ≥ 3,000/mcL
* Absolute Neutrophil Count (ANC) ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
* Creatinine ≤ 2.0 mg/dl Or Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* The patient must express HLA class I allele HLA-A*0201 for NY-ESO-1/LAGE.
* Patient must have proven positive tumor sample for NY-ESO-1 as determined by an H score for immunohistochemistry staining. Positive expression is defined as an H score ≥ 100 where the H score = [2 x (% cells 2+) + 3 x (% cells 3+)].

NOTE: The percentages of negative or weakly stained nuclei (i.e. 1+) are not to be included in the calculation of the H score.

* Female subjects of childbearing potential must have a negative pregnancy test and both male and female (of childbearing potential) subjects must agree to use reliable methods of contraception during the study.
* Ability of the patient (or legally authorized representative if applicable) to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients who have had 2 or more regimens containing cytotoxic chemotherapy for metastatic melanoma.
* Patients may not be receiving any other investigational agents.
* Patients with active brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide or other agents used in the study.
* Active infection
* Prior malignancy (except non-melanoma skin cancer) within 3 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. All patients will undergo a cardiac stress test for evaluation of cardiac function.
* Pregnant or nursing females
* Active infection with HIV, HBV or HCV as defined below, due to the immunosuppressive effects of cyclophosphamide used and the unknown risks associated with viral replication.
* Positive serology for HIV
* Active Hepatitis B infection as determined by test for hepatitis B surface antigen.
* Active Hepatitis C. Patients will be screened for HCV antibody. If the HCV antibody is positive, a screening HCV RNA by any RT-PCR or bDNA assay must be performed at screening by a local laboratory with a CLIA certification or its equivalent. Eligibility will be determined based on a negative screening value. The test is not required if documentation of a negative result of a HCV RNA test performed within 60 days prior to screening is provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald P Linette, MD, PhD, Principal Investigator — Washington University School of Medicine; Harriet Kluger, MD, Principal Investigator — Yale New Haven Hospital
Locations (2):
- United States (2):
  - Yale School of Medicine, New Haven, Connecticut
  - Washington University in St. Louis, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days: Participants who received cytoreductive chemotherapy followed by infusion of lentivirus-mediated genetically engineered NY-ESO-1ᶜ²⁵⁹T (Target dose: 5-10 billion cells)
Period: Overall Study
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 49 [41 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Related to Study Treatment
Description: Number of Participants with NCI CTC V.4 Adverse Events related to study treatment greater than or equal to Grade 3
Time Frame: Up to 12 months
Population: Participants who received cytoreductive chemotherapy followed by IV infusion of NY-ESO-1ᶜ²⁵⁹T
Measure: Count of Participants; unit: Participants
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days
Number analyzed (Participants) | 4
Participants | 3

2. Secondary Outcome: Tumor Response
Description: Number of participants with response as assessed by RECIST (version 1.1) criteria.
Time Frame: Change from Baseline, every 4 weeks until Month 5 and then every other month through Month 11
Measure: Count of Participants; unit: Participants
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: Determine the Functional Properties and Phenotype of Modified T-cells From Peripheral Blood and Tumor Sites.
Description: Measurement of functionality of NY-ESO-1ᶜ²⁵⁹T cells in the blood and tumor sites.
Time Frame: 8 Weeks post T-cell infusion
Population: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T with functionality data
Measure: Number; unit: percentage of T cell sub population
Units Other Than Participants: T-cell sub population
Groups:
- Subject 1 - Manufactured Product: Participants who received cytoreductive chemotherapy followed by infusion of lentivirus-mediated genetically engineered NY-ESO-1ᶜ²⁵⁹T (Target dose: 5-10 billion cells)
Arm/Group | Subject 1 - Manufactured Product | Subject 1 - Day 60 | Subject 2 - Manufactured Product | Subject 2 - Day 60
Number analyzed (Participants) | 1 | 1 | 1 | 1
Number analyzed (T-cell sub population) | 7 | 7 | 7 | 7
percentage of T cell sub population
  %Stem Cell Memory | 31.1354 | 61.545 | 18.65934 | 6.9
  %Central Memory | 14.62221 | 3.42 | 6.85214 | 6.9
  %Effector Memory RA | 36.329 | 32.475 | 34.50644 | 82.7
  %Effector Memory | 17.8215 | 2.56 | 39.99068 | 3.45
  %LAG-3+ | 0.40391 | 0 | 1.23488 | 0
  %PD-1+ | 1.24694 | 0.855 | 4.11214 | 0
  %TIM-3+ | 97.74411 | 5.985 | 95.2126 | 10.35

4. Secondary Outcome: Peak Persistence of Modified T-cells in the Peripheral Blood
Description: Measurement of NY-ESO-1ᶜ²⁵⁹T cells in blood (copies of WPRE per µg of genomic PBMC DNA)
Time Frame: Days 1, 5-9, 12-16, weekly thereafter through Week 12, monthly thereafter through Month 12, and during LTFU
Population: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T with persistence data
Measure: Mean (Full Range); unit: copies per μg of DNA
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days
Number analyzed (Participants) | 4
copies per μg of DNA | 56561.22 [24984.1 to 126679]

ADVERSE EVENTS:
Time Frame: Start of lymphodepletion to end of intervention phase (up to 12 months post T-cell infusion)
Description: Participants who received NY-ESO-1ᶜ²⁵⁹T
Arm/Group | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (4)
Pyrexia (General disorders) | 1 (4)
Platelet count decreased (Investigations) | 1 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYESO-1ᶜ²⁵⁹T Cells Administered IV as a Split Dose Over 2 Days (N=4)
Fatigue (General disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Neutropenia decreased (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less